CLINICAL TRIAL: NCT04194385
Title: Comparison of Perioperative Analgesic Efficacy of Ultrasonography Guided Upper Trunk Block and Costoclavicular Infraclavicular Brachial Plexus Block in Arthroscopic Shoulder Surgery
Brief Title: Upper Trunk Block Versus Costoclavicular Block For Arthroscopic Shoulder Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 71306642-050-05-04-
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Shoulder Pain; Phrenic Nerve Paralysis
Keywords: bupivacaine; costoclavicular block; upper trunk block
MeSH Terms: conditions — Shoulder Pain | interventions — Cervical Plexus Block

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Upper trunk block (Active Comparator): In the supraclavicular region, UTB will be applied with 20 ml % 0.25 bupivacaine with 5 mcg/ml epinephrine.
  Interventions: Procedure: Upper trunk block; Procedure: Diaphragmatic function assessment; Procedure: Cervical plexus blockade
- Costoclavicular brachial plexus block (Active Comparator): In the infraclavicular region, CCBPB will be applied with 20 ml % 0.25 bupivacaine with 5 mcg/ml epinephrine.
  Interventions: Procedure: Costoclavicular block; Procedure: Diaphragmatic function assessment; Procedure: Cervical plexus blockade

INTERVENTIONS:
Procedure: Upper trunk block — Block will be applied to supraclavicular zone by 20 ml % 0.25 bupivacaine with 5 mcg/ml epinephrine .
  Other Names: Upper trunk brachial plexus block
  Arms: Upper trunk block
Procedure: Costoclavicular block — Block will be applied to infraclavicular zone by 20 ml % 0.25 bupivacaine with 5 mcg/ml epinephrine.
  Other Names: Costoclavicular brachial plexus block
  Arms: Costoclavicular brachial plexus block
Procedure: Diaphragmatic function assessment — Diaphragmatic excursion will be assessed under ultrasound immediately before and after regional anesthesia.
  Other Names: Detection of diaphragmatic paralysis with ultrasound guidance
Procedure: Cervical plexus blockade — Block will be applied at thyroid cartilage level via 10 ml % 0.25 bupivacaine.
  Other Names: Superficial cervical plexus blockade

SUMMARY:
Interscalene brachial plexus block is known as the gold standard for analgesia after shoulder surgery, but limits the use of ipsilateral phrenic nerve paralysis. Recently, interest in potential diaphragm-sparing alternative blocks has increased for patients undergoing shoulder surgery.Two of these blocks are upper trunk block (UTB) and costoclavicular brachial plexus (CCBPB) block. This randomized controlled trial will compare ultrasound-guided UTB and CCBPB in patients undergoing arthroscopic shoulder surgery.

The main outcome is pain intensity score at 30 minutes after arrival in the post anesthesia care unit (PACU) as measured by a numerical rating scale (NRS) from 0 to 10. The investigators research hypothesis is that UTB and CCBPB will result in equivalent postoperative analgesia at 30 minutes in the PACU.

ELIGIBILITY:
Inclusion Criteria:

1. American Association of Anesthesiologists (ASA) physical status I - III
2. BMI 20 to 35 kg / m2
3. Patients scheduled for elective arthroscopic shoulder surgery

Exclusion Criteria:

1. Patients who refuse to participate in the study,
2. Pre-existing (obstructive or restrictive) lung disease,
3. Coagulopathy,
4. Sepsis,
5. Hepatic or renal insufficiency,
6. Pregnancy
7. Allergy to local anesthetic drugs,
8. Chronic pain condition requiring opioid intake at home,
9. Surgery in the neck or infraclavicular region
10. BMI above 40.
11. History of psychiatric diseases needing treatment.
12. Failure of nerve block performed in the preoperative block room
13. Substance abuse history

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-05-10 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Detection of diaphragmatic paralysis by ultrasonography | 30 minutes after block application
  Ipsilateral diaphragmatic excursion 30 minutes after block completion

SECONDARY OUTCOMES:
Postoperative opioid consumption | 24 hour after surgery
  Total amount of tramadol consumption during the first 24 hours after surgery. Patient controlled analgesia to be inserted.
Pain intensity score | 30 minutes, 1,3, 6, 12, 24 hour after surgery
  Postoperative pain assessed with verbal rating scale (VRS 0: no pain 10:pain as bad as can be )
Block perform time | The time from the needle enters the skin until the block is completed
  Block application time will be recorded
Block onset time | Until sensory and motor block occurs
  Block onset time will be evaluated and recorded.
Intraoperative fentanyl requirement | From the beginning to the end of the operation
  During the operation, 0.5 μg/kg fentanyl was administered to the patient in case of a 20% increase in the mean blood pressure and heart rate compared to the baseline values
Patient satisfaction: NRS | 24 hour after surgery
  Patient satisfaction measured using a NRS 0 to 10 (0 = unsatisfied; 10 =very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Serdar Yeşiltaş, Instructor, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Fatih, Turkey (Türkiye)